CLINICAL TRIAL: NCT00381316
Title: Comparison of Diagnostic Rest/Stress SPECT Results for Patients With Myocardial Ischemia and Infarction Using Myoview in Both Single and Dual Isotope Acquisition Approaches
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: GE Healthcare (Industry)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 143-002
Record Dates: First submitted 2006-09-25; First posted 2006-09-27 (Estimated); Last update posted 2007-12-05 (Estimated); Status verified 2007-11

CONDITIONS: Coronary Artery Disease
MeSH Terms: conditions — Coronary Artery Disease

ARMS (2):
- 1 (Active Comparator): Thallous Chloride T1-201
  Interventions: Drug: Thallous Chloride T1-201
- 2 (Active Comparator): Technetium Tc99m Tetrofosmin injections
  Interventions: Drug: Technetium Tc99m Tetrofosmin injections

INTERVENTIONS:
Drug: Technetium Tc99m Tetrofosmin injections — Single Isotope: be 555 to 888 MBq (15 to 24 mCi) MYOVIEW at Rest/i.v./bolus.
  Arms: 2
Drug: Thallous Chloride T1-201 — Myoview SPECT Imaging
  Arms: 1

SUMMARY:
The study is designed to determine whether a dual isotope protocol is equivalent to a single isotope in the diagnosis of myocardial ischemia and infarction using MYOVIEW SPECT imaging.

ELIGIBILITY:
Inclusion Criteria:

1. The subject is 18 years old or older.
2. Male subjects or non-lactating female subjects, who are either surgically sterile (has had a documented bilateral oophorectomy and/or documented hysterectomy), postmenopausal (cessation of menses for more than 1 year), or for women of childbearing potential, the results of a serum or urine human chorionic gonadotropin pregnancy test, performed at screening within 24 hours before dosing (with the result known before investigational medicinal product administration) must be negative.
3. The subject is able and willing to comply with study procedures (i.e., 1 SPECT imaging at Stress, 2 SPECT imagings at Rest) and signed and dated informed consent is obtained.
4. The subject is suspected of or known of having CAD based on the subject's clinical signs, symptoms, or examinations .
5. The subject is referred for Rest/Stress (exercise or pharmacological) MPS-SPECT for known or suspected CAD (as clinically required).

Exclusion Criteria:

1. The subject was previously included in this study.
2. The subject received an IMP within 30 days before or is scheduled to receive one during or in the next 30 days after IMP administration.
3. The subject has known allergies to any product used in this study or its constituents, including subjects who are not able to exercise and have contraindications to Adenosine (e.g., Asthmatics).
4. The subject presents any clinically active, serious, life-threatening disease, with a life expectancy of less than 1 month.
5. The subject has no contraindications to any of the study procedures (e.g. physical exercise) or the involved drugs (Myoview, Thallium-201, Adenosine or Dipyridamole) such as e.g. 2nd or 3rd degree AV-block, SS syndrome, bradycardia, bronchoconstrictive or bronchospastic lung disease.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 291 (Actual)
Dates: Start 2006-07; Study Completion 2006-12 (Actual)

PRIMARY OUTCOMES:
The diagnostic results ("normal" versus "abnormal") of the dual-isotope and single isotope myocardial SPECT examinations will be compared for equivalence on a subject level for the Uninformed and Informed Analysis Groups.

CONTACTS AND LOCATIONS:
Overall Officials: Andre Mueller-York, Study Director — GE Healthcare
Locations (1):
- GE Healthcare, Princeton, New Jersey, United States